CLINICAL TRIAL: NCT00598143
Title: Biomarkers of Molecular Risk in Smokers
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Weill Medical College of Cornell University (Other); Vanderbilt University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 04-141
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Surveys and Questionnaires; Urine Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva Samples

GROUPS / COHORTS (2):
- Group A: Ten healthy smokers will provide a saliva sample used to genotype UGT1A7 and complete a questionnaire to assess understanding of and willingness to participate in molecular risk assessments.
  Interventions: Behavioral: Vignette, questionnaires and Saliva Samples
- Group B: Thirty smokers will receive standard smoking cessation therapy and provide urine specimens for PGE-M analysis at approximate 3-monthly intervals over one year. Self-reported smoking status and expired-air carbon monoxide (CO) will also be recorded at 3-monthly clinic visits.
  Interventions: Behavioral: Urine Collection, Smoking cessation treatment

INTERVENTIONS:
Behavioral: Vignette, questionnaires and Saliva Samples — The short vignette discusses the health implications of potential molecular markers of cancer risk assessment. The questionnaire asks several multiple-choice questions to assess the participant's interest in and understanding of molecular risk assessment. Patients are instructed to swish with 10cc of Scope mouthwash and to expectorate into a sterile 50cc conical tube.
  Groups: Group A
Behavioral: Urine Collection, Smoking cessation treatment — Single void urine specimens (approximately 50 ml) will be collected in pre-labeled specimen containers on a 3-monthly (±1 month) basis for 12 months. Standard evidence-based therapy for smoking cessation, including behavioral therapy and pharmacological therapy, is provided.
  Groups: Group B

SUMMARY:
Doctors at MSKCC are doing this research study to see if smokers are interested in the idea that genes might be markers of cancer risk, and to see if smokers would want to learn this information about their risk if it were available.

Different versions of the gene called UGT1A7 are found in different people. Certain versions of this gene can increase the risk of cancer in people. In this study, doctors will determine the different types of UGT1A7 in smokers and find out whether smokers show good interest and understanding. The information from this study will be used in future studies to identify smokers at increased risk for cancer, and to help smokers quit.

DETAILED DESCRIPTION:
This study consists of two arms; both of which are observational studies of molecular assessments of risk for tobacco related cancer. Arm A of the protocol is a pilot crosssectional study that evaluates the feasibility of obtaining and testing a genetic marker of cancer susceptibility (UGT1A7 polymorphisms) in smokers. It also explores smokers' interest in and comprehension of genetic risk assessments as possible tools for increasing motivation for smoking cessation. The second arm of this protocol, Arm B, is an observational prospective evaluation of a putative noninvasive biomarker of tobacco smoke exposure - urinary prostaglandin E-metabolite (PGE-M) - in smokers motivated to reduce and/or cease smoking.

ELIGIBILITY:
Inclusion Criteria:

* Arm A
* 18 years or older;
* >5 packyear history of smoking;
* Ability to understand and sign informed consent.
* Arm B
* 18 years or older;
* >10 packyear history of smoking;
* Intention to taper and/or quit smoking within 6 months
* Ability to understand and sign informed consent.

Exclusion Criteria:

* Arm A
* Diagnosis of any cancer in the preceding twelve months; (excluding non melanoma skin cancer).
* Arm B
* Diagnosis of any cancer in the preceding twelve months; (excluding non melanoma skin cancer).
* Use of any COX-2 inhibitor, steroid, or non-steroidal anti-inflammatory medication (excluding cardioprotective aspirin > 81mg/d) within one week of urine collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: MSKCC clinics
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2005-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Estimate accrual rates and smokers' willingness to provide saliva for cancer risk assessment. | conclusion of study

SECONDARY OUTCOMES:
Evaluate the effect of smoking reduction and/or cessation on levels of urinary PGE-M. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Jay Boyle, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org